CLINICAL TRIAL: NCT05061979
Title: Open-label, Single-dose Study to Evaluate the Pharmacokinetics and Safety of BAY1747846 in Participants With Impaired Renal Function in Comparison to Matched Participants With Normal Renal Function
Brief Title: A Study to Evaluate the Pharmacokinetics (How it Moves Into, Through and Out From the Body) of a New Gadolinium-based Contrast Agent (GBCA) After Injection and How Safe it is in Participants With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21180
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Contrast Enhancement in Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mild renal impairment (Experimental): Participants with mild renal impairment will receive a single dose of BAY1747846.
  Interventions: Drug: BAY1747846
- Moderate renal impairment (Experimental): Participants with moderate renal impairment will receive a single dose of BAY1747846.
  Interventions: Drug: BAY1747846
- Normal renal function (Experimental): Participants with normal renal function will receive a single dose of BAY1747846.
  Interventions: Drug: BAY1747846

INTERVENTIONS:
Drug: BAY1747846 — Solution for intravenous (IV) injection, single dose

SUMMARY:
Researchers in this study want to learn how a new contrast agent for magnetic resonance imaging (MRI) called BAY1747846 moves into, through and out of the body (pharmacokinetics) after injection in participants with normal and impaired renal function. Impaired renal function is a condition where the kidneys do not work as well as they should.

BAY1747846 belongs to the class gadolinium-based contrast agents (GBCAs). The way the body removes GBCAs including BAY1747846 from the blood is through the kidneys. So, when the kidneys are not working normally, it takes longer to remove BAY1747846 out of the body.

The participants in this study will either have normal renal function, or will have mild or moderate impaired renal function. The participants will receive BAY1747846 one time through a needle into a vein.

During the study, the participants will visit the study site about 6 times. The participants will stay at the study site for up to 9 days. Each participant will be in the study for up to 7 months. During the study, the doctors will:

* check the participants' overall health
* take blood and urine samples
* ask the participants about what medications they are taking and what adverse events they are having An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 79 years of age inclusive, at the time of signing the informed consent
* Renally Impaired Participants and Disease Characteristics

  * Mildly or moderately decreased renal function, as assessed by estimated glomerular filtration rate (eGFR). Mildly impaired renal function: eGFR: 60 up to 89 mL/min/1.73 m^2 (inclusive); Moderately impaired renal function: eGFR: 30 up to 59 mL/min/1.73 m^2 (inclusive)
  * Stable renal disease, i.e. a serum creatinine value determined 3 or more months before screening (e.g. during routine diagnostics) should not differ by more than 25% from the serum creatinine value determined at screening
* Participants with normal renal function: Normal renal function, as assessed by eGFR ≥90 mL/min/1.73 m^2
* Body mass index (BMI) within the range 18 - 40 kg/m^2 (inclusive)
* Body weight (bw) ≥ 45 kg
* Study participants of reproductive potential must agree to use adequate contraception when sexually active.
* Male participants must agree not to donate sperm from the signing of the ICF until the follow-up visit on Day 12 (± 2d).

Exclusion Criteria:

* Any relevant disease (other than those related to renal impairment for the renal impaired participants) within 4 weeks prior to study drug administration including infections and acute gastro-intestinal diseases (vomiting, diarrhea, constipation) requiring medical treatment
* Acute renal failure or acute nephritis within the past 2 years
* Febrile illness within 1 week before study drug administration
* Malignancy diagnosed or treated within the past 5 years (hepatocellular carcinoma within the past 2 years). This does not include adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin
* Conditions associated with a risk of hypersensitivity reactions as judged by the investigator
* Any participant not able to produce urine and/or needing dialysis
* Dialysis for acute renal failure within the previous 6 months prior to administration of study intervention
* Contrast agent administration within one month prior to screening or during the screening period
* Indication for immunosuppressants, receiving cytotoxic therapy, immunosuppressive therapy, or other immunotherapy within 6 months prior to administration of study intervention
* Clinically relevant abnormalities in physical examination, ECG, clinical chemistry, hematology, or urinalysis as judged by the investigator
* Heart rate below 45 bpm or above 110 bpm
* Systolic blood pressure below 90 mmHg or above 170 mmHg
* Diastolic blood pressure below 45 or above 105 mmHg
* Indication or evidence for long QT syndrome for all participants; additionally for participants with normal renal function: QT interval corrected using Fridericia's method (QTcF) > 470 msec
* History of COVID-19 within 6 months prior to screening
* Long COVID-19 syndrome or other clinically relevant COVID-19-related symptoms or sequela
* Incomplete SARS-CoV-2 vaccination
* Vaccination planned before completion of the last study visit

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve from zero to infinity of BAY1747846 after single dose administration (AUC) | Pre-dose until 7 days post-dose
Maximum observed drug concentration of BAY1747846 in plasma after single dose administration (Cmax) | Pre-dose until 7 days post-dose
Total body clearance of BAY1747846 normalized by body weight | Pre-dose until 7 days post-dose

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events | After administration of study intervention up to Day 12 (± 2 days)
Number of participants with treatment-emergent adverse events categorized by severity | After administration of study intervention up to Day 12 (± 2 days)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Alliance for Multispecialty Research, LLC - Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Fadini T, Sutter G, Klein S, Busemann E, Vendel E, Vis P, Heitmeier S, Frenzel T, Ebert W, Hofmann BM. Pharmacokinetics, Safety, and Dialyzability of Gadoquatrane in Patients With Impaired Renal Function: A Comprehensive Investigation Using Clinical Trial Data, Modeling and Simulation, and In Vitro Data. Invest Radiol. 2025 Nov 1;60(11):779-790. doi: 10.1097/RLI.0000000000001191. PMID 40215351
- [Derived] Lohrke J, Berger M, Frenzel T, Hilger CS, Jost G, Panknin O, Bauser M, Ebert W, Pietsch H. Preclinical Profile of Gadoquatrane: A Novel Tetrameric, Macrocyclic High Relaxivity Gadolinium-Based Contrast Agent. Invest Radiol. 2022 Oct 1;57(10):629-638. doi: 10.1097/RLI.0000000000000889. Epub 2022 Jun 13. PMID 35703267